CLINICAL TRIAL: NCT04050917
Title: Development of Wearable Stimulation App to Increase Hand Functional Recovery in Patients With Neurologic Movement
Brief Title: Smartwatch App for Vibration Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: MUSC Foundation for Research Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00088976
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Physical Disability
Keywords: physical stimulation; Subliminal stimulation; stroke rehabilitation; upper extremity; paresis; hand function; occupational therapy; physical therapy
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real stimulation (Experimental): The smartwatch produces vibration stimulation.
  Interventions: Device: real stimulation
- No stimulation (Sham Comparator): The smartwatch produces no vibration.
  Interventions: Device: no stimulation

INTERVENTIONS:
Device: real stimulation — The smartwatch generates imperceptible vibratory stimulation.
  Arms: Real stimulation
Device: no stimulation — The smartwatch generates no stimulation.
  Arms: No stimulation

SUMMARY:
The objective of this study is to determine if the acute effect of vibration from a smartwatch on hand function is comparable to the effect of an existing laboratory prototype.

DETAILED DESCRIPTION:
More than 4 million stroke survivors in the U.S. suffer from post-stroke hand disability. As hands are our primary means of interacting with the world, post-stroke hand impairment diminishes stroke survivors' abilities for activities of daily living including self-care, hygiene, employment, and leisure, and lowers independence. Hand impairment is difficult to treat. Limited resources in rehabilitation services and financial burdens make it impractical to simply increase rehabilitation service visits within the current healthcare system.

One way to augment hand function recovery is peripheral sensory stimulation. Afferent input is a powerful driver of change in the motor cortex. Sensory stimulation has been shown to improve motor recovery in previous studies. In particular, promising preliminary results have been obtained by using imperceptible random-frequency vibration applied via a watch. However, the laboratory prototype device for delivering this vibration must be improved in the form factor for patient adoption.

Therefore, we developed an App that can be installed in smartwatches and control the vibrator within the smartwatch to deliver vibratory stimulation to the user. The objective of this study is to determine if the acute effect of vibration from a smartwatch on hand function is comparable to the effect of an existing laboratory prototype.

ELIGIBILITY:
Inclusion Criteria:

* Age = 18 or older
* At least 6 months post stroke
* The ability to perform The Box and Block Test with a score greater than zero and less than 40.

Exclusion Criteria:

* Rigidity (Modified Ashworth Scale=5)
* Complete upper limb deafferentation
* Comorbidity (peripheral neuropathy, orthopaedic conditions in the hand that limit ranges of motion, premorbid neurologic conditions, compromised skin integrity of the hand/wrist due to long-term use of blood thinners)
* Language barrier or cognitive impairment that precludes following instructions and/or providing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | 20 minute
  number of blocks moved

SECONDARY OUTCOMES:
Nine Hole Peg Test | 20 minute
  time it takes to complete the test

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Caorlina, Charleston, South Carolina, United States